CLINICAL TRIAL: NCT06012188
Title: The Effect of Sleeping Companion Toy Given to Earthquake Victims Aged 3-6 on Children's Sleeping Habits
Brief Title: Aged 3-6 on Children's Sleeping Habits
Acronym: [Sleep]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, Elif Simay KOÇ, Lecturer, Kilis 7 Aralik University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Kilis7AralikU_E_S_KOÇ00
Record Dates: First submitted 2023-08-21; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Sleep Habits; Child

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Children in the experimental group will be given a sleeping companion toy.
  Interventions: Other: sleep toy
- Control group (No Intervention): No intervention will be made on the control group.

INTERVENTIONS:
Other: sleep toy — The parents of the children in the experimental group will be given a sleeping companion toy to present to their children. At the end of 15 days, the Children's Sleep Habits scale will be applied as a post-test to evaluate the effect of the sleep companion toy.
  Arms: Experimental group

SUMMARY:
One of the most important points in sleep health is the sleep habits of children. Natural disasters cause sleep problems in children, increase or decrease in sleep duration, change in sleep habits and adversely affect sleep quality. According to Erikson's theory of psychosocial development, children aged 3-6 are entrepreneurs. It is the period when children begin to learn and apply the rules, and independence efforts are developed in the child. Negative sleep behaviors and sleep problems are common during this period, but children can develop positive sleep habits if properly and consistently guided by their parents. Rituals such as fairy tales, lullabies, night lamps, toys can help children relax and calm down and gain sleep habits.

DETAILED DESCRIPTION:
The research design is a randomized controlled experimental type study designed to evaluate the effect of sleeping companion toys given to earthquake survivors aged 3-6 years on children's sleep habits.The Children's Sleep Habits Scale will be used to determine the sleep habits of children in the earthquake area by pre-interviewing the parents of children aged 3-6. Children aged 3-6 with sleep problems will be divided into control and experimental groups according to their scale scores. The part up to this section constitutes the preliminary test of our research.

Children aged 3-6 years in the control group and their parents will not receive any intervention.

Families of the children in the experimental group will be given a sleep companion gift to give to their children. Children's sleep habits scale will be applied as a post-test to determine children's sleep problems 15 days after they receive a gift from their sleep friend. Then, sleep habits scale mean scores will be calculated and a comparison will be made between pretest and posttest mean scores.

ELIGIBILITY:
Inclusion Criteria:

* Ages ranging from 3 to 6
* Earthquake living
* Parents being literate
* Parents and children who accepted the study and gave voluntary consent

Exclusion Criteria:

* Being a 3-6 year old child who has previously had a sleep disorder finding
* Being visually, hearing or speech impaired
* Children aged 3-6 with mental disorders

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-08-30 (Estimated); Primary Completion 2023-09-13 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Children's Sleep Habits Scale | 15 day
  The Children's Sleep Habits Scale will be used to determine children's sleep habits and sleep-related problems. Children's Sleep Habits Scale consists of 8 sub-dimensions and a total of 33 items.In grading the scale, parents are asked to respond as 1=rarely (0-1 times a week), 2=sometimes (2-4 times a week), and 3=usually (5-7 times a week). A minimum of 33 points and a maximum of 99 points are taken from the scale. The total test score is obtained by summing the scores obtained from the items one by one.
  It is accepted that those who have a total score of 41 and above with CIAS have clinical sleep problems.

CONTACTS AND LOCATIONS:
Overall Officials: FATMA KURUDİREK, Principal Investigator — fsaban@atauni.edu.tr; Türkan KADİROĞLU, Principal Investigator — t.kadiroglu@atauni.edu.tr

IPD SHARING:
Plan to Share IPD: No